CLINICAL TRIAL: NCT05863598
Title: A Randomized Controlled Trial of an Interactive Non-Stigmatizing Intervention to Prevent Eating Disorders in Youths Through Strengthening of Protective Factors
Brief Title: Prevention of Eating Disorders Through Optimization of Protective Factors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Uppsala University (Other); Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Ata Ghaderi, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-01039
Record Dates: First submitted 2023-04-28; First posted 2023-05-18 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-10

CONDITIONS: Body Dissatisfaction; Eating Disorders
Keywords: eating disorders; body dissatisfaction; risk factors; buffering factors; incidence; efficacy; cost-effectiveness
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: This is randomized controlled trials. Participants will be randomized to the active prevention program, or to a placebo (expressive writing). The intervention is brief (four weeks only). Recruitment of the participants (n=644) will take one year (anticipated)After the intervention, they will receive a booster session and will be followed up every 6 months, for 36 months post-intervention.
Who Masked: Outcomes Assessor
Masking Description: Randomization will be conducted using a randomization list. As soon as a participant is eligible after providing baseline data and a clinical interview, the assessment staff will ask the coordinator to check what condition the participant should be assigned to based on the randomization list. The participants will be informed. At follow-ups, the assessors will not be aware of the intervention condition of each participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhancing protective factors (Experimental): Participants will learn to improve their body image through body appreciation tasks, body image flexibility and focus on body functionality appreciation. They also learn to focus on important life values, be more accepting of themselves, and learn to eat regularly and with attention to bodily needs and signals. This is don in interactive ways, and by using a cognitive dissonance frame.
  Interventions: Behavioral: Enhancing protective factors
- Expressive writing (Placebo Comparator): Participants will be instructed to write about any thoughts, feelings, images, memories, interceptions, ideas or emotions related to their body for the same during as the active intervention (i.e., 40 minutes/week across four consecutive weeks).
  Interventions: Behavioral: Expressive writing

INTERVENTIONS:
Behavioral: Enhancing protective factors — Participants will watch some short movies and infographics, and will be asked to argue for the importance of body image flexibility, body functionality appreciation, etc.
  Arms: Enhancing protective factors
Behavioral: Expressive writing — Participants will reflect and write about any cognitions or emotions they can have in relation to their bodies.
  Arms: Expressive writing

SUMMARY:
The goal of thin randomized controlled trial is to investigate the efficacy of a prevention program for reducing the incidence of eating disorders among youth (15-20). We target youth at these ages who experience a subjective sense of body dissatisfaction, and are thus at increased risk of developing an eating disorder.

The prevention program is based on improving protective factors such as body appreciation, body image flexibility, intuitive eating, and acceptance. It will be compared to a credible placebo (expressive writing).

DETAILED DESCRIPTION:
Research area and aims:

Eating disorders (EDs) are common and cause significant morbidity and mortality. Due to stigma, only 25% seek help and only 50% fully recover after receiving treatments. Large-scale prevention is urgently needed to reduce the emergence and burden of EDs at a population level. However, current prevention programs do not meet requirements for efficient and economically attractive large-scale implementation. The main aim of this project is to investigate the efficacy and cost-effectiveness of a scalable, brief, and interactive prevention program based on reinforcement of protective factors against EDs using a randomized controlled design. A focus on protective factors disrupts the processes by which risk factors increase the probability for EDs to emerge and minimizes the risks for stigmatization.

Research questions:

1. How effective is an internet-based prevention program, that reinforces protective factors against EDs, in reducing the onset of EDs 6, 12, 24, and 36 months post-intervention?
2. Does the intervention reduce the incidence of EDs through enhancement of specifically targeted protective factors (mediators)?
3. Is prevention of EDs based on reinforcement of protective factors cost-effective?
4. How do the participant experience their participation in these two interventions?

Other research questions concern gender differences in enrollment and compliance, potential moderators of outcome, participation in booster sessions, and potential risk for stigma.

ELIGIBILITY:
Inclusion Criteria: Youth and young people (15-20 years) with a subjective experience of body dissatisfaction.

Exclusion Criteria: Indications of depression, or suicidality, as well as presence of an eating disorder, or other conditions that may require medical attention, or conditions that makes it impossible to complete the intervention (e.g., not being able to read and write in Swedish).

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 644 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of eating disorders through the Eating disorders examination (EDE) (Fairburn, 2008, Guilford Press). | Baseline to 36 months post-intervention
  The Eating disorders examination interview is the gold standard to establish diagnoses of eating disorders and will be used at baseline and to investigate the incidence of eating disorders (ED) during the follow-up period (36 months post intervention). Diagnostic status will be specified based on specific criteria for each ED diagnosis.

SECONDARY OUTCOMES:
Change in body dissatisfaction through the Body Shape questionnaire: BSQ (Welch et al, 2011: Beh Res Ther, 49, 85-91). | From baseline, up to 36 months post-intervention
  The Body Shape questionnaire (Brief version: 8 items) measures body dissatisfaction. It has good psychometric properties. Items are scored on a Likert-type scale from 1 (Never) to 6 (Always). Higher scores indicate more body dissatisfaction.
Change in drive for muscularity through the Drive for Muscularity Scale (DMS: McCreary& Sasse, 2000, J Am Coll Health, 48, 297-304). | From baseline, up to 36 months post-intervention
  The Drive for Muscularity Scale (15 items) measures one of the risk factors for ED. It has good psychometrics. Items are rated on a scale from 1 to 6. Higher scores indicate stronger drive for muscularity.
Change in the internalization of thin ideal through the Ideal Body Stereotype Scale-Revised (IBSS-R: Stice et al, 2008, J Consult Clin Pschol, 76, 329-340) | From baseline, up to 36 months post-intervention
  The Body Stereotype Scale-Revised (6 items) measures the internalization of the current thinness ideal, which is a risk factors for ED. It has good psychometrics. Items are rated on a scale from 1 to 5. Higher scores indicate more internalization of the thin ideal.
Change in quality of life through The Brunnsviken Quality of Life Scale (BBQ: Lindner et al, 2016, Cogn Behav Ther, 45, 182-195). | From baseline, up to 36 months post-intervention
  The Brunnsviken Quality of Life Scale is a brief instrument (12 items) developed in Sweden with good psychometrics to measure quality of life. The items are rated on a scale from 0 to 4. Higher scores indicate stronger satisfaction with life.
Change in body appreciation through the Body Appreciation Scale (BAS: Tylka & Wood-Bacalow, 2015, Body Image, 12, 53-67). | From baseline, up to 36 months post-intervention
  The Body Appreciation Scale (10 items) has good psychometrics. The items are scored on a scale from 1 to 5. Higher scores indicate more body appreciation.
Change in body functionality appreciation through the Functionality Appreciation Scale (FAS: Alleva et al, 2017, Body Image, 23, 28-44). | From baseline, up to 36 months post-intervention
  The Functionality Appreciation Scale (7 items) has good psychometrics. Items are rated on a scale from 1 to 5. Higher scores indicate higher appreciation of body functionality.
Change in body image flexibility through the Body Image Acceptance and Action Questionnaire (BI-AAQ-5: Sandoz et al, 2013, J Cont Behav Science, 2, 39-48). | From baseline, up to 36 months post-intervention
  The Body Image Acceptance and Action Questionnaire measures body image flexibility (5 items), which is another protective factor. Items are rated on a scale from 1 to 7. Higher scores indicate more body image flexibility.
Change in intuitive eating through the Intuitive Eating Scale (IES: Tylka & Kroon Van Diest, 2013, J Cons Psychol, 60,137-153). | From baseline, up to 36 months post-intervention
  The Intuitive Eating Scale (23 items) is an established measure of intuitive eating. It has good psychometric properties. Items are rated on a scale from 1 to 5. Higher scores indicate more intuitive eating.
Change in self-compassion through the Self-Compassion Scale (SCS: Raes et al., 2011, Clin Psychol Psychother, 18, 250-255). | From baseline, up to 36 months post-intervention
  The Self-Compassion Scale (Brief version: 12 items) has good psychometrics. It provides information on an important protective factor. Items are rated on a scale from 1 to 5. Higher scores indicate higher self-compassion.
Change in life values through the Bull's-Eye Values Survey (BE-VS: Lundgren et al, 2012, Cogn Behav Pract, 19, 518-526). | From baseline, up to 36 months post-intervention
  The Bull's-Eye Values Survey helps to ascertain what ares in life (i.e., personal values) seem important to each participant. It has been adapted by providing the instructions through a brief instructional video instead of lengthy text. The importance of life directions are rated on a scale from 0 to 7. Higher scores indicate more importance. The proximity to life values is rated on a scale from 1 to 7. Higher scores indicate more proximity, where 7 is the bull's eye.

OTHER OUTCOMES:
Moderators of outcomes: Sex, Age, Socio-economic status. | Baseline assessment
  Data on sex (Male or Female), age (15-20) and socioeconomic status (level of education) will be used to investigate whether they moderated the rate of enrollment, compliance (how many modules of the program they complete), and outcome.
Experience of stigma and iatrogenic effects through the Self-reported risk of stigma and iatrogenic effect | Post-intervention (i.e., 5 weeks after the start of intervention)
  Any experience of stigma or iatrogenic effects related to the intervention/study will be investigated through specifically designed questions for the study
Experience of stigma and iatrogenic effects through the Self-reported risk of stigma and iatrogenic effect. | 6-months post-intervention
  Any experience of stigma or iatrogenic effects related to the intervention/study will be investigated through specifically designed questions for the study.
Experience of stigma and iatrogenic effects through the Self-reported risk of stigma and iatrogenic effect. | 12-months post-intervention
  Any experience of stigma or iatrogenic effects related to the intervention/study will be investigated through specifically designed questions for the study.
Experience of stigma and iatrogenic effects through the Self-reported risk of stigma and iatrogenic effect. | 24-months post-intervention
  Any experience of stigma or iatrogenic effects related to the intervention/study will be investigated through specifically designed questions for the study.
Experience of stigma and iatrogenic effects through the Self-reported risk of stigma and iatrogenic effect. | 36-months post-intervention
  Any experience of stigma or iatrogenic effects related to the intervention/study will be investigated through specifically designed questions for the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ata Ghaderi, PhD, Principal Investigator — PI employed at Karolinska Institutet
Locations (1):
- Karolinska Institutet, Solna, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghaderi A, Stice E, Andersson G, Eno Persson J, Allzen E. A randomized controlled trial of the effectiveness of virtually delivered Body Project (vBP) groups to prevent eating disorders. J Consult Clin Psychol. 2020 Jul;88(7):643-656. doi: 10.1037/ccp0000506. PMID 32551736
- [Background] Andrew R, Tiggemann M, Clark L. The protective role of body appreciation against media-induced body dissatisfaction. Body Image. 2015 Sep;15:98-104. doi: 10.1016/j.bodyim.2015.07.005. Epub 2015 Aug 24. PMID 26311661
- [Background] Atkinson MJ, Wade TD. Mindfulness-based prevention for eating disorders: A school-based cluster randomized controlled study. Int J Eat Disord. 2015 Nov;48(7):1024-37. doi: 10.1002/eat.22416. Epub 2015 Jun 6. PMID 26052831
- [Background] Burychka D, Miragall M, Banos RM. Towards a Comprehensive Understanding of Body Image: Integrating Positive Body Image, Embodiment and Self-Compassion. Psychol Belg. 2021 Jul 27;61(1):248-261. doi: 10.5334/pb.1057. eCollection 2021. PMID 34394951
- [Background] Homan KJ, Tylka TL. Self-compassion moderates body comparison and appearance self-worth's inverse relationships with body appreciation. Body Image. 2015 Sep;15:1-7. doi: 10.1016/j.bodyim.2015.04.007. Epub 2015 May 16. PMID 25978272
- [Background] Levine MP, Smolak L. The role of protective factors in the prevention of negative body image and disordered eating. Eat Disord. 2016;24(1):39-46. doi: 10.1080/10640266.2015.1113826. Epub 2015 Dec 7. No abstract available. PMID 26643272
- [Background] Linardon J, Tylka TL, Fuller-Tyszkiewicz M. Intuitive eating and its psychological correlates: A meta-analysis. Int J Eat Disord. 2021 Jul;54(7):1073-1098. doi: 10.1002/eat.23509. Epub 2021 Mar 30. PMID 33786858
- [Background] Mensinger JL, Granche JL, Cox SA, Henretty JR. Sexual and gender minority individuals report higher rates of abuse and more severe eating disorder symptoms than cisgender heterosexual individuals at admission to eating disorder treatment. Int J Eat Disord. 2020 Apr;53(4):541-554. doi: 10.1002/eat.23257. Epub 2020 Mar 13. PMID 32167198
- [Background] Moffitt RL, Neumann DL, Williamson SP. Comparing the efficacy of a brief self-esteem and self-compassion intervention for state body dissatisfaction and self-improvement motivation. Body Image. 2018 Dec;27:67-76. doi: 10.1016/j.bodyim.2018.08.008. Epub 2018 Aug 23. PMID 30144731
- [Background] Ahlen J, Hursti T, Tanner L, Tokay Z, Ghaderi A. Prevention of Anxiety and Depression in Swedish School Children: a Cluster-Randomized Effectiveness Study. Prev Sci. 2018 Feb;19(2):147-158. doi: 10.1007/s11121-017-0821-1. PMID 28730396
- [Background] Koller KA, Thompson KA, Miller AJ, Walsh EC, Bardone-Cone AM. Body appreciation and intuitive eating in eating disorder recovery. Int J Eat Disord. 2020 Aug;53(8):1261-1269. doi: 10.1002/eat.23238. Epub 2020 Feb 5. PMID 32020677